CLINICAL TRIAL: NCT02127879
Title: High-frequency Repetitive Transcranial Magnetic Stimulation for Negative Symptoms in Schizophrenia: The Double-blind Sham-controlled Study
Brief Title: Intensive Transcranial Magnetic Stimulation for Negative Symptoms in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Tomáš Svěrák, Mgr., Masaryk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TSRPMMLA1; 61300 (Other: Department of Psychiatry, Faculty of Medicine, Masaryk University, Brno, Czech Republic)
Record Dates: First submitted 2014-04-26; First posted 2014-05-01 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: Repetitive Transcranial Magnetic Stimulation; Schizophrenia; Negative symptoms; Intensive; Transcranial Magnetic Stimulation, Repetitive
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): Active Treatment 10 Hz rTMS of left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimulation with sham coil (Sham Comparator): Sham coil Treatment 10 Hz rTMS of left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Transcranial Magnetic Stimulation with sham coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — 16 sessions/4 days (4 sessions per day), 2000 stimuli per one session, 20 trains per session (train interval= 10 sec., intertrain interval= 30sec.), stimulation intensity 110 % related to the individual resting motor threshold; in total 32,000 stimuli, 20 min. pause is between every stimulation session for safety reasons.v
  Other Names: Magstim Rapid 2
  Arms: Transcranial Magnetic Stimulation
Device: Transcranial Magnetic Stimulation with sham coil — 16 sessions/4 days (4 sessions per day), 2000 stimuli per one session, 20 trains per session (train interval= 10 sec., intertrain interval= 30sec.), stimulation intensity 110 % related to the individual resting motor threshold; in total 32,000 stimuli, 20 min. Pause is between every stimulation session for safety reasons.
  Other Names: Magstim Rapid 2 with sham coil
  Arms: Transcranial Magnetic Stimulation with sham coil

SUMMARY:
The main purpose of this study is to determine whether intensive repetitive transcranial magnetic stimulation (I-rTMS) is effective in the treatment of negative symptoms in schizophrenia patients and whether it has a positive influence on their cognitive functions, social functions, quality of life, alpha frequency and cortical silent period changes. Also, this study should provide data about safety and tolerability this I-rTMS treatment in schizophrenia patients.

DETAILED DESCRIPTION:
Patients undergo 5x EEG from safety and research reasons during the study. Stimulation coil location (left DLPFC) is determined by magnetic resonance imaging (1,5T, 3D- TFE, voxel size 1 x 1 x 1 mm, Intera MR scanner) and stereotactic neuronavigation (Brainsight Frameless).

Patients are evaluated by several psychiatric scales. Positive and negative symptom scale (PANSS) is applied before the first stimulation, at the end of every stimulation day and two weeks after the last stimulation (a total 6). Other psychiatric evaluations used are Clinical global impression (CGI), Sheehan disability scale (SDS), Personal and social performance scale (PSP) and Montgomery-Asberg Depression Scale (MADRS), Calgary depression scale for schizophrenia (CDSS); (MADRS and CDSS are for the exclusion of depression). These scales were used only before the start of the first stimulation, after its completion and two weeks after the last test.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent, the patient must be able and willing to participate in a research study,
* Undergo an examination by international neuropsychiatric questionnaire MINI - PLUS to confirm the diagnosis of schizophrenia
* schizophrenic illness duration longer than one year,
* have a stable and consistent drug treatment at least two weeks prior the rTMS treatment
* persistent negative symptoms without further psychiatric comorbidity (like depression, mania, anxiety disorders, personality disorders, etc.) in the foreground of the illness
* The sum of negative scores in the range Positive and negative symptom score (PANSS) must be 20 points or higher and at least one item from the area of negative symptoms (N1-N7) must be ≥ 4 points (at least moderate, clinically significant symptoms),
* improvement in negative symptom-sum (measuring by PANSS) must be 10% or lower during the last two weeks before rTMS stimulation.

Exclusion Criteria:

* involuntary stay in a psychiatric clinic during the recruitment of patients;
* clinically relevant unstable medical conditions;
* factors incompatible with the use of rTMS, such as pacemakers, heart pumps and other metal implants;
* history of epileptic seizures or the presence of epileptic activity documented on the basis of EEG
* current treatment with anticonvulsant acting drugs such as anticonvulsants, benzodiazepines (10mg/D or less of diazepam or equivalent dosage of other benzodiazepines);
* lack of cognitive skills for participation;
* clinically relevant psychiatric comorbidity (any other axis 1 diagnosis) detected using MINI Plus, including the current abuse of drugs and alcohol;
* heart attack or traumatic head injury in the anamnesis
* Patient unable to undergo a brain MRI
* Acute risk of suicide;
* knowledge of Czech language at a level that does not allow fill the required test battery;
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in negative symptoms measured by Negative scale in Positive and Negative Syndrome Scale (PANSS) | Baseline, Week 3

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 5 weeks
  Patients undergoing five times EEG during the study for safety reasons. The researcher assigns patients on their health and mental condition by Visual Analogous Scale every day before and after rTMS stimulation.

OTHER OUTCOMES:
Change from baseline in quality of life in the Quality of Life questionaire (SQUALA) at week 3 | At baseline, Week 3
Change from baseline in cognitive functions measured by Verbal learning test, Rey- Osterrieth complex figure, D2 test, Repeating numbers memory test, London tower test, Verbal fluency test at week 3 | Baseline, Week 3
  Verbal learning test testing memory (based on Rey Auditory Verbal Learning Test), Rey- Osterrieth complex figure testing testing sensomotoric and visuospatial skills, D2 test testing attention, Repeating numbers memory test testing working memory, London Tower test testing executive functions and Verbal fluency test testing verbal fluency and recalling of words
Change from baseline in social functions measured by Sheehan Disability Scale (SDS) and by Personal and Social Performance Scale (PSP) at week 3 | Baseline, Week 3
Change from baseline in global clinical improvement measured by Clinical Global Impression (CGI) at week 3 | Baseline, Week 3
Change from baseline in alpha frequency measured by EEG at week 3 | Baseline, Week 3
Change from baseline in cortical silent period measured by transcranial magnetic stimulation at week 3 | Baseline, Week 3

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Svěrák, Mgr., Principal Investigator — Brno University Hospital; Radovan Přikryl, Prof., Study Director — Brno University Hospital
Locations (1):
- Departement of psychiatry, University Hospital, Brno, Czech Republic, Czechia